CLINICAL TRIAL: NCT02223091
Title: Prospective, Multi-center, Cluster-randomized, Pragmatic, Mixed-method Pilot Study Evaluating a Consultation Training Program for Physicians Within the Framework of KOKON (Competence Network Complementary Medicine in Oncology)
Brief Title: KOKON Consultation on Complementary Medicine in Oncology - a Pilot Study
Acronym: KOKON-AS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. Claudia M. Witt, MBA, Charite University, Berlin, Germany
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: KOKON-109863
Record Dates: First submitted 2014-07-02; First posted 2014-08-22 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Breast-cancer
Keywords: complementary therapies; consultants; medical oncology; breast-cancer; education
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Consultation by a trained physician (Experimental): The physicians of this group receive a free consultation training program on skills regarding consultations on complementary medicine for breast-cancer patients. The training was developed by a multi-professional team and is comprised of three parts: (1) online-training, (2) on-site-training, and (3) consultation manual. Each of the physicians will counsel 10 patients. The patients in this group therefore receive a consultation by a trained physician.
  Interventions: Behavioral: Consultation by a trained physician
- Consultation by an untrained physician (Active Comparator): The physicians of the control arm receive no training. Each will counsel 10 patients. The patients in this group therefore receive a consultation by an untrained physician.
  Interventions: Behavioral: Consultation by an untrained physician

INTERVENTIONS:
Behavioral: Consultation by a trained physician
  Arms: Consultation by a trained physician
Behavioral: Consultation by an untrained physician
  Arms: Consultation by an untrained physician

SUMMARY:
The aim of the study is to investigate the effect of a consultation training program for physicians on the quality of their consultations of breast cancer patients regarding complementary medicine. We assume that the training program might enhance the communication of relevant information, empathy of the physicians or satisfaction with the consultation.

ELIGIBILITY:
Inclusion Criteria for physicians:

* age >18 years
* working in a breast center of comprehensive cancer center
* able to consult 10 patients within working hours
* training group: able to participate in on-site-training
* not primarily treating the patients that are consulted
* good language skills (for consultations)
* informed consent

Inclusion Criteria for patients:

* age > 18 years
* female
* diagnosis of breast-cancer
* patient in the participating center
* good language skills (for consultations)
* informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-09; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the training program | day 1-7
  This is an exploratory study. The main aim is to evaluate the effectiveness of the training program which will be achieved using the different outcome measures defined here as secondary outcome measures.

SECONDARY OUTCOMES:
Knowledge about complementary medicine in oncology and consultations (physicians) | day 1-7
  Questions regarding different topics relating to complementary medicine in oncology and consultations of oncology patients
Evaluation of each consultation session (physicians) | day 1-7
  Evaluation of the consultation session by the physicians (e.g. time spent on the consultation, difficulties, empathy etc.)
Empathy: CARE (patient) | day 1-7
  Empathy is assessed via an adaption of the German version of the Consultation and Relational Empathy scale (CARE)
Empathy: REM (patient) | day 1-7
  Empathy is assessed via an adapted version of the Rating Scales for the Assessment of Empathic Communication in Medical Interviews (REM)
Satisfaction with the consultation session (patient) | day 1-7
  Satisfaction with the consultation session is assessed via questions developed by the study team.
Quality of information (patient) | day 1-7
  Quality of the information is assessed via questions developed by the study team
Qualitative analysis of focus groups (physicians) | day 1-7
  Focus groups will be conducted with each group of physicians (trained and untrained). They will be analyzed using qualitative methods.
Qualitative analysis of videotapings of consultation sessions | day 1-7
  In each group (consulations by trained and by untrained physicians) 8 consultation sessions will be videotaped and analyzed with qualitative methods.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Witt, MD, MBA, Principal Investigator — Charite University, Berlin, Germany
Locations (8):
- Germany (8):
  - Brustzentrum am Vivantes Klinikum am Urban, Berlin
  - Brustzentrum im Sana-Klinikum Lichtenberg, Berlin
  - Brustzentrum, Klinik für Gynäkologie, Charité, Campus Mitte, Berlin
  - DRK Kliniken Westend, Brustzentrum, Berlin
  - Universitätsklinikum Heidelberg, Brustzentrum, Heidelberg
  - Brustzentrum der LMU München, München
  - Brustzentrum Klinikum Nürnberg-Nord, Nuremberg
  - Universitätsklinikum Würzburg, Frauenklinik und Poliklinik, Würzburg

REFERENCES:
- [Derived] Blodt S, Mittring N, Schutzler L, Fischer F, Holmberg C, Horneber M, Stapf A, Witt CM. A consultation training program for physicians for communication about complementary medicine with breast cancer patients: a prospective, multi-center, cluster-randomized, mixed-method pilot study. BMC Cancer. 2016 Nov 4;16(1):843. doi: 10.1186/s12885-016-2884-y. PMID 27809814